CLINICAL TRIAL: NCT02650232
Title: Pilot Study to Evaluate the Somnotouch Device to Quantify Spontaneous Baroreflex Sensitivity in Healthy Subjects and in Patients With Heart Failure
Brief Title: Pilot Study to Evaluate the Somnotouch Device to Quantify Spontaneous Baroreflex Sensitivity
Acronym: SOMNO-BRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: LivaNova (Industry); SomnoMedics (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 15-A01215-44
Record Dates: First submitted 2015-12-21; First posted 2016-01-08 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Healthy; Heart Failure
Keywords: Volunteers
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Young Healthy Volunteers (Other): We will evaluate in this group (18 - 40 y) the use of the SOMNOtouch system to quantify the spontaneous baroreflex sensitivity
  Interventions: Device: SOMNOtouch device (Somnomedics); Procedure: Orthostatic test; Device: Finapres Nova device (FMS system)
- Old Healthy Volunteers (Other): We will evaluate in this group (50 - 80 y) the use of the SOMNOtouch system to quantify the spontaneous baroreflex sensitivity
  Interventions: Device: SOMNOtouch device (Somnomedics); Procedure: Orthostatic test; Device: Finapres Nova device (FMS system)
- Patients with heart failure (Other): We will evaluate in this group (50 - 80 y + Heart failure) the use of the SOMNOtouch system to quantify the spontaneous baroreflex sensitivity
  Interventions: Device: SOMNOtouch device (Somnomedics); Procedure: Orthostatic test; Device: Finapres Nova device (FMS system)

INTERVENTIONS:
Device: SOMNOtouch device (Somnomedics) — In each arm, we will evaluate the capacity of SOMNOtouch to measure the baroreflex sensitivity compared to Finapre Nova (reference)
Procedure: Orthostatic test — For each arm we will proceed to an orthostatic test day one and day two with :
  * 10 minutes in supine position
  * 10 minutes in sitting position
  * 5 minutes in standing position
  * 5 minutes in supine position
Device: Finapres Nova device (FMS system)

SUMMARY:
To measure the spontaneous baroreflex sensitivity in ambulatory patient, a device made for measuring blood pressure beat by beat and continuously, the SOMNOtouch system, could be a useful tool. The SOMNOtouch system has never been used to assess the sensitivity of the baroreflex. A good correlation for measuring the baroreflex sensitivity between the system "SOMNOtouch" and digital photoplethysmography as a reference method is expected but should be evaluated. The main purpuse is to evaluate the SOMNOtouch system to quantify the spontaneous baroreflex sensitivity in healthy young subjects, in elderly healthy subjects and in subjects with heart failure. We will also evaluate the feasibility of measuring the baroreflex sensitivity in ambulatory conditions for 24 hours, the variations in sensitivity of the baroreflex sensitivity between day and night, the reproducibility of orthostatic tolerance test.

ELIGIBILITY:
For healthy volunteers

Inclusion Criteria:

* good health
* normal ECG
* cardiac ejection fraction > 50%

Exclusion Criteria:

* with chronic disease or treatment
* under law protection
* not affiliated to the national health insurance

For patients with heart failure

Inclusion Criteria:

* clinically sable
* with sinusal heart rhythm
* without sign of neuropathy
* cardiac ejection fraction < 50%

Exclusion Criteria:

* with pace maker
* under law protection
* not affiliated to the national health insurance
* skin lesion or severe allergia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Coefficient of correlation in baroreflex sensitivity measurements between SOMNOTOUCH and FINAPRES nova during the orthostatic test | Day one
  baroreflex sensitivity is measured by comparison of the variations in heart rate and in blood pressure (baroreflexe slope method & fransfer function method). We will compare this baroreflex sensitivity obtained from SOMNOTOUCH measurement and from Finapres nova measurements (coefficient of correlation)

SECONDARY OUTCOMES:
Coefficient of correlation in baroreflex sensitivity measurements between day one and day two during the orthostatic test | Day two vs Day one
  baroreflex sensitivity is measured by comparison of the variations in heart rate and in blood pressure (baroreflex slope method & fransfer function method). We will compare this baroreflex sensitivity between the two active orthostatic tests (coefficient of correlation).
Duration of recordings in hours over 24 hours that allows the measurement of the spontaneous baroreflex sensitivity with the SOMNOTOUCH system | Day one (24 hours)
  We will mesure over 24 hours the duration in hours when the measurement of the baroreflex sensitivity is possible taken in account the quality of the physiological signals.
Difference in the baroreflex sensitivity between Day & Night | Day one (24 hours)
  We will compare the baroreflex sensitivity between day and night in each group and between groups.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU d'Angers, Angers, Maine Et Loire
  - CH de Cholet, Cholet, Maine Et Loire